CLINICAL TRIAL: NCT00005381
Title: Prevalence of Sleep Apnea in Women
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Edward Bixler, Principal Investigator, Milton S. Hershey Medical Center
Other Study IDs: 4286; R01HL051931 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Lung Diseases; Sleep Apnea Syndromes
MeSH Terms: conditions — Lung Diseases; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify the prevalence of sleep apnea (SA) in women and its relationship to age; to predict those women at risk for sleep apnea; and to define the natural history of those with sleep apnea.

DETAILED DESCRIPTION:
BACKGROUND:

Often sleep apnea is accompanied by considerable morbidity; the associated excessive daytime sleepiness, cardiovascular abnormalities and cognitive impairment impact greatly on daytime functioning. The obese, hypertensives, elderly and postmenopausal women are reported to be at increased risk for sleep apnea. The investigators published on the prevalence of sleep apnea in several special populations: elderly subjects without sleep complaints and insomniac, narcoleptic, hypertensive and obese patients. They established the prevalence of sleep apnea in men based on the sleep laboratory evaluation of approximately 1,000 men randomly selected from a randomly generated telephone sample of 4,364 men from the general population. Their preliminary estimate of prevalence was that about 2.2 percent of the adult male population have clinically diagnosable sleep apnea. Further, in the male sample, the age distribution was not linearly related to age. Rather, it peaked at approximately age 55. Finally, the major risk factors appeared to be obesity and snoring. The differences in the male/female ratio in clinical and selected populations ranged from 10.0:1 to 1.9:1. One recent study suggested that the prevalence of sleep apnea in women was about two-fold less than in men. However, this study did not sample the general population and used only a restricted age range (30 to 60 years) which did not allow the assessment of the influence of menopause. Thus, the prevalence of sleep apnea in women in the general population remained largely undetermined.

DESIGN NARRATIVE:

In order to establish the prevalence in women with reasonable precision, the prevalence study employed a two-stage sample modified from the prevalence study in men in the following two ways: an expanded telephone sample (N=12,219 women) selected randomly from the general population was evaluated, for clinically relevant risk factors for sleep apnea; and 2) a second sample (N=1,000) selected randomly from the first sample based on higher risk for sleep apnea (including the additional risk factor of menopause) was evaluated in the sleep laboratory to determine the presence of sleep apnea. This strategy yielded an adequate power in order to establish the prevalence of sleep apnea requiring treatment and sleep disordered breathing in women in the general population as well as result in a large enough sample to establish the association between risk factors and sleep apnea in women. In order to perform gender analyses, the study compared previously published data from a total of 4,364 men interviewed in an expanded telephone sample and 741men evaluated in the sleep laboratory.

ELIGIBILITY:
Stratified random sample based on risk severity obtained during phone interview

Ages: 20 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stratified random sample following initial phone survey
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 1995-10-29 (Actual); Primary Completion 1998-08-02 (Actual); Study Completion 1998-08-02 (Actual)

PRIMARY OUTCOMES:
Sleep Disordered Breathing | Immediately upon time of recording
  Apnea/hypopnea index

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bixler EO, Vgontzas AN, Lin HM, Ten Have T, Rein J, Vela-Bueno A, Kales A. Prevalence of sleep-disordered breathing in women: effects of gender. Am J Respir Crit Care Med. 2001 Mar;163(3 Pt 1):608-13. doi: 10.1164/ajrccm.163.3.9911064. PMID 11254512